CLINICAL TRIAL: NCT06851364
Title: Efficacy of 0.38% and 0.18% Sodium Hyaluronate Ocular Lubricants for Dry Eye: A Randomized Trial in Adult Gazan Participants
Brief Title: Efficacy of 0.38% and 0.18% Sodium Hyaluronate Ocular Lubricants for Dry Eye in Adult Gazan Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Islamic University of Gaza, Gaza, Palestine (Unknown)
Responsible Party: Principal Investigator, Mohd Zulfaezal Che Azemin, Professor, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC/HC/883/21
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye
Keywords: Evaporative Dry Eye (EDE); Ocular Surface Disease; Tear Film Dysfunction; Ocular Lubricants
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.38% Sodium Hyaluronate (SH) Eye Drops (Experimental)
  Interventions: Drug: 0.38% Sodium Hyaluronate (SH) Eye Drops
- 0.18% Sodium Hyaluronate (SH) Eye Drops (Experimental)
  Interventions: Drug: 0.18% Sodium Hyaluronate Eye Drops
- Normal Saline Eye Drops (Placebo Comparator)
  Interventions: Drug: Normal Saline Eye Drops

INTERVENTIONS:
Drug: 0.38% Sodium Hyaluronate (SH) Eye Drops — A lubricant eye drop containing 0.38% sodium hyaluronate (SH), designed to improve tear film stability and ocular surface health in individuals with moderate to severe dry eye disease (DED).
  The formulation has a higher viscosity and retention time, potentially offering better symptom relief for evaporative dry eye (EDE).
  Arms: 0.38% Sodium Hyaluronate (SH) Eye Drops
Drug: 0.18% Sodium Hyaluronate Eye Drops — A lubricant eye drop containing 0.18% sodium hyaluronate (SH), used to alleviate dry eye symptoms and improve tear film stability.
  This formulation has a lower viscosity compared to 0.38% SH, potentially providing faster absorption but with shorter ocular surface retention.
  Arms: 0.18% Sodium Hyaluronate (SH) Eye Drops
Drug: Normal Saline Eye Drops — A non-active control treatment consisting of sterile normal saline (0.9% NaCl) used as a placebo comparator.
  It provides temporary moisture but lacks the viscoelastic and therapeutic properties of sodium hyaluronate.
  Arms: Normal Saline Eye Drops

SUMMARY:
The goal of this completed clinical trial was to determine if 0.38% and 0.18% sodium hyaluronate (SH) lubricant eye drops improve symptoms of moderate to severe dry eye disease (DED) in adult Gazan participants. The main questions it aimed to answer were:

1. Did 0.38% and 0.18% SH eye drops improve Arab-Ocular Surface Disease Index (Arab-OSDI) scores?
2. Did these eye drops improve tear break-up time (TBUT), corneal fluorescein staining (CFS), and lissamine green conjunctival staining (LGS)?
3. Did 0.38% SH provide greater benefits in evaporative dry eye (EDE) compared to 0.18% SH and normal saline?
4. Researchers compared 0.38% SH, 0.18% SH, and normal saline eye drops to evaluate their effectiveness in symptom relief and clinical improvements.

Participants:

1. Applied their assigned eye drops three times daily for six weeks Used normal saline eye drops for the first week before starting their assigned treatment
2. Underwent clinical assessments at weeks 1, 3, and 6, including Arab-OSDI scoring, TBUT, CFS, and LGS tests
3. The study began on October 30, 2022, and was completed on February 3, 2023, with 45 participants each completing a 6-week trial period.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 40 years.
* Residents of South Gaza Strip.
* Diagnosed with moderate to severe dry eye disease (DED) based on Arab-OSDI score (≥ 23).

Exclusion Criteria:

* History of systemic diseases (e.g., rheumatoid arthritis, Sjögren syndrome, thyroid disorders).
* Previous punctal plugs or punctal cautery treatment for ocular surface pathologies.
* Presence of pterygium, evident lid/orbital disease with lagophthalmos, or history of punctal cautery.
* Contact lens (CL) users who always need to wear CLs.
* History of ocular surgeries within 6 months or LASIK within 12 months.
* Use of medications that could affect study results (e.g., antihistamines, antidepressants, aspirin, anticholinergics, corticosteroids) or recent use of central nervous system or hormonal medications within 30 days.
* Current use of ocular medications or those planning to start new medications during the study.
* Pregnant participants or those with ocular pathologies beyond DED and refractive errors.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Arab-OSDI Score from baseline (Visit 2) to week 6 (Visit 5) | 6 weeks
  The primary outcome is the improvement in dry eye symptoms, as measured by the Arabic version of the Ocular Surface Disease Index (Arab-OSDI) questionnaire. A reduction in the Arab-OSDI score indicates symptom improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic University of Gaza (IUG), Gaza, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
The study investigators may share individual participant data (IPD) upon reasonable request, in compliance with ethical and legal requirements. Data will be shared in a de-identified format to protect participant privacy. Access to the data will require approval from the research team and may be granted for purposes of meta-analyses or further research related to dry eye disease.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form) will be available starting 6 months after publication of primary results. The data will remain accessible for 5 years from the release date or upon reasonable request from qualified researchers.
Access Criteria: Qualified researchers affiliated with academic institutions, research organizations, or healthcare entities may request access to the Individual Participant Data (IPD) and supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form). Access will be granted upon submission of a research proposal outlining the intended use of the data, along with institutional ethics approval or data-use agreements, if applicable. Requests will be reviewed by the study's data-sharing committee, and approved researchers will be provided access via a secure data-sharing platform. Data will be shared in a de-identified format to protect participant confidentiality, in compliance with ethical and regulatory guidelines.
URL: https://scholar.google.com/citations?user=Lv0N40sAAAAJ&hl=en